CLINICAL TRIAL: NCT05924828
Title: Comparison of sTREM-1, sTREM-2, Presepsin, and Its Association With Periodontitis: A Randomized Controlled Three-Blinded Clinic Study
Brief Title: sTREM-1, sTREM-2, Presepsin, and Periodontitis
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Didem OZKAL EMINOGLU, assistant professor, Ataturk University
Other Study IDs: atauniperio3
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: periodontitis; sTREM-1; sTREM-2; Presepsin
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: participants without periodontitis
  Interventions: Other: no intervention
- periodontitis: participants with stage-3 periodontitis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention
  Other Names: periodontitis; healthy

SUMMARY:
The goal of this observational study is to compare saliva sTREM-1, sTREM-2, Presepsin levels and sTREM-1/sTREM-2 ratio of participants with/without periodontitis.

The main question it aims to answer is there a relationship between saliva sTREM-1, sTREM-2, Presepsin levels, sTREM-1/sTREM-2 ratio and periodontitis.

Participants will give saliva samples without any intervention

DETAILED DESCRIPTION:
Periodontitis is a chronic, inflammatory disease with a cyclical course with active and passive periods, which may result in the destruction of gingival fibers, resorption of alveolar bone, and subsequent tooth loss, by spreading the inflammatory event that started in the gingiva to the tissues supporting the tooth as a result of the effects of bacteria. The disease is closely associated with many systemic conditions. These conditions include diabetes, cardiovascular diseases, respiratory diseases, birth complications, pregnancy, puberty.

sTREM-1, the soluble form of TREM-1 resulting from the cleavage by MMP (matrix metalloproteinase) of the extracellular portion of this receptor, was identified in 2004. Higher concentrations of sTREM-1 were noted in gingival crevicular fluid (GCF) and saliva from patients with periodontitis and correlated with certain periodontal clinical parameters (Plaque Index [PlI], Gingival Index [GI], PPD or clinical attachment loss [CAL]). TREM-2, another member of the TREM family, is also synthesised by macrophages and together with its receptor, DNAX-activating protein of 12 kDa (DAP12), functions to suppress the proinflammatory response. Initial studies with TREM-2 in microglia cells showed that it plays an important role in suppressing TNF-α and IL-6 levels. The secretion of presepsin has been reported as a stimulus of monocytes phagocytosis. Therefore, recognition of presepsin is predictable even in healthy non-infective individuals. The concept for presepsin proposes that its levels should be measureable in non-infective individuals, increase the early steps of bacterial infections, and its levels should be dependent on the intensity of the innate immune induction.

The study material will be 70 adult individuals who applied to Atatürk University Faculty of Dentistry, Department of Periodontology for different reasons {1. group (H): periodontally healthy individuals, group 2 (P): individuals with periodontitis}. Saliva samples will be collected from the participants without any periodontal intervention. sTREM-1, sTREM-2, Presepsin levels will be studied.

The aim of this study; to evaluate the saliva sTREM-1, sTREM-2, Presepsin levels and sTREM-1/sTREM-2 ratio in the saliva samples of patients with periodontitis by comparing them with healthy controls, and to investigate the association in the pathogenesis of periodontitis or a simple marker of disease activity in the light of these findings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals should not have any systemic disease that may or may not require medication, including salivary gland pathologies, and not particularly thyroid organ pathologies.
* Individuals have not been continuously treated with anti-inflammatory, antioxidant or similar drugs in the last 6 months,
* Individuals have not received periodontal treatment until 6 months ago,
* Individuals must have at least 14 teeth
* Patients diagnosed with stage 3 periodontitis

Exclusion Criteria:

* Having a systemic disease such as cardiovascular, diabetes, hypertension, thyroid organ pathologies, chronic kidney failure
* Being pregnant/breastfeeding
* Being on medication for any reason
* Being a smoker/tobacco user
* Having another periodontal disease other than periodontitis
* Having a chronic inflammatory disease (COPD, asthma)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals who referred to Atatürk University, Department of Periodontology
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
sTREM-1, sTREM-2, Presepsin | 0-1 hours of the diagnosis
  sTREM-1, sTREM-2, Presepsin levels in saliva

CONTACTS AND LOCATIONS:
Overall Officials: DİDEM ÖZKAL EMİNOĞLU, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided